CLINICAL TRIAL: NCT01237262
Title: Evaluation of Lymphocytic Infiltrate, Dendritic Cells and Cytokines Expression in Psoriatic Lesion and Normal Skin Before and After Adalimumab Therapy
Brief Title: Evaluation of Lymphocytic Infiltrate, Dendritic Cells and Cytokines Expression in Psoriatic Lesion and Normal Skin Before and After TNF Alfa Inhibitors Therapy
Acronym: ELIDACE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Padova (Other)
Responsible Party: ANDREA PESERICO, University of Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ELIDACE in PSO
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Moderate to Severe Psoriasis.; Absolute Number, Density of Immune Infiltrate and Dendritic Cells and Inflammatory Cytokines Expression Pattern.
Keywords: psoriasis; immune infiltrate; dendritic cells; cytokine expression
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab; Etanercept; Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TNF alfa inhibitors (Active Comparator): Male and female adult patients with a diagnosis of moderate to severe psoriasis (when PASI score is > 10 and BSA is > 10%). The overall study enrolment plan is 20 patients. Patients will be screened before the beginning of clinical trial by blood sample in order to exclude major contraindications to use of anti TNF α drugs.
  Interventions: Drug: Adalimumab, etanercept, infliximab

INTERVENTIONS:
Drug: Adalimumab, etanercept, infliximab — Adalimumab at a dose of 80 mg at week 0 (Baseline) and successively 40 mg every other week starting from week1 and up to week 15. Adalimumab will be administered as subcutaneous injection.
  Etanercept at a dose of 50 mg every week, as subcutaneous injection. Infliximab at a dose of 5 mg/kg at week 0 (Baseline), then at week 2 and every 8 weeks.

SUMMARY:
The efficacy of TNF alfa inhibitors in the treatment of psoriasis has been documented in many studies.

Their effect on dendritic cells has been scarcely studied. TNF- α has a central role in dendritic cell biology, both for their maturity and mobilization of peripheral tissues to secondary lymphoid organs.

The primary objectives of this study are:

* To document absolute number, density of immune infiltrate and dendritic cells and inflammatory cytokines expression pattern (particularly IFN α and IL-32) in psoriasic lesions vs normal skin of the same patient
* To describe changes in such cell numbers and expression patterns upon 16 weeks treatment with TNF alfa inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects > 18 years of age, affected by moderate to severe psoriasis
* Subject has had clinical diagnosis of psoriasis for at least 12 months, stable plaque psoriasis for at least 2 months before screening (subjects with concurrent psoriatic arthritis may be enrolled).
* Subject is naıve to TNF-antagonist therapy and efalizumab.
* Subjects are considered eligible according to the following tuberculosis screening criteria:

  1. Have no history of latent or active TB prior to screening;
  2. Have no signs or symptoms suggestive of active TB upon medical history and/or physical examination;
  3. Within 1 month prior to the first administration of study medication, have negative diagnostic tuberculin skin test.
* Normal chest X-ray within 3 months prior to screening with no evidence of malignancy, infection, current or old TB.
* Subjects' screening and baseline clinical data must be within the normal limit, including the results of medical history, physical examination and laboratory evaluation (complete blood count, serum values for liver enzymes, bilirubin, glucose, albumin, creatinine and urine analysis).
* Willing and able to comply with the protocol requirements for the duration of the study.
* Women of childbearing potential must be using adequate birth control measure throughout the study and for 150 days (5 months) after study completion.

Exclusion Criteria:

* Pregnant or breast-feeding women, or women who are planning pregnancy.
* Patients not suitable for TNF alfa inhibitors therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-11; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
changes in absolute numbers, density of immunocompetent cells and inflammatory cytokines expression pattern in psoriasic lesions vs normal skin of the same patient, pre and post-TNF alfa inhibitors treatment. | 12 months
  * To document absolute number, density of immune infiltrate and dendritic cells and inflammatory cytokines expression pattern (particularly IFN α and IL-32) in psoriasic lesions vs normal skin of the same patient
  * To describe changes in such cell numbers and expression patterns upon 16 weeks treatment with biologics.

CONTACTS AND LOCATIONS:
Overall Officials: ANDREA PESERICO, PROF, Study Chair — University of Padova
Locations (1):
- Stefano Piaserico, Padua, Italy, Italy

REFERENCES:
- [Background] Nestle FO, Kaplan DH, Barker J. Psoriasis. N Engl J Med. 2009 Jul 30;361(5):496-509. doi: 10.1056/NEJMra0804595. No abstract available. PMID 19641206
- [Background] Bedini C, Nasorri F, Girolomoni G, Pita Od, Cavani A. Antitumour necrosis factor-alpha chimeric antibody (infliximab) inhibits activation of skin-homing CD4+ and CD8+ T lymphocytes and impairs dendritic cell function. Br J Dermatol. 2007 Aug;157(2):249-58. doi: 10.1111/j.1365-2133.2007.07945.x. Epub 2007 May 8. PMID 17489975